CLINICAL TRIAL: NCT01060371
Title: Clinical Research Consortium for Spinocerebellar Ataxias (CRC-SCA) to Study Natural History Study of and Genetic Modifiers in Spinocerebellar Ataxias (SCA)
Brief Title: Natural History Study of and Genetic Modifiers in Spinocerebellar Ataxias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florida (Other)
Collaborators: National Ataxia Foundation (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201700740; 505-2009 (Other: Legacy study); OCR16458 (Other: Universiy of Florida); NCT01223417 (obsolete NCT alias)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 3; Spinocerebellar Ataxia Type 6
Keywords: Spinocerebellar Ataxia; Natural History; Genetic Modifiers; DNA testing
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collection for DNA analysis and genetic modifier study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Spinocerebellar Ataxia 1: If you decide to participate in this study, the following study procedures will be performed:
  * blood collection for DNA testing, analysis (genetic modifier study) and banking
  * Medical history
  * Physical exam
  * Scale for Assessment and Rating of Ataxia (SARA)
  * Timed measure of your hand dexterity and walking (25 ft)
  * Questionnaire about your daily living activities, your physical and mental quality of life and assessment of depression.
  * Disease stage estimation by the clinician.
  * Demographics and disease-related information (i.e. age, sex, race, age at disease onset, disease duration)
  * Review of your medical records
  Interventions: Genetic: All Participants
- Spinocerebellar Ataxia 2: If you decide to participate in this study, the following study procedures will be performed:
  * blood collection for DNA testing, analysis (genetic modifier study) and banking
  * Medical history
  * Physical exam
  * Scale for Assessment and Rating of Ataxia (SARA)
  * Timed measure of your hand dexterity and walking (25 ft)
  * Questionnaire about your daily living activities, your physical and mental quality of life and assessment of depression.
  * Disease stage estimation by the clinician.
  * Demographics and disease-related information (i.e. age, sex, race, age at disease onset, disease duration)
  * Review of your medical records
  Interventions: Genetic: All Participants
- Spinocerebellar Ataxia 3: If you decide to participate in this study, the following study procedures will be performed:
  * blood collection for DNA testing, analysis (genetic modifier study) and banking
  * Medical history
  * Physical exam
  * Scale for Assessment and Rating of Ataxia (SARA)
  * Timed measure of your hand dexterity and walking (25 ft)
  * Questionnaire about your daily living activities, your physical and mental quality of life and assessment of depression.
  * Disease stage estimation by the clinician.
  * Demographics and disease-related information (i.e. age, sex, race, age at disease onset, disease duration)
  * Review of your medical records
  Interventions: Genetic: All Participants
- Spinocerebellar Ataxia 6: If you decide to participate in this study, the following study procedures will be performed:
  * blood collection for DNA testing, analysis (genetic modifier study) and banking
  * Medical history
  * Physical exam
  * Scale for Assessment and Rating of Ataxia (SARA)
  * Timed measure of your hand dexterity and walking (25 ft)
  * Questionnaire about your daily living activities, your physical and mental quality of life and assessment of depression.
  * Disease stage estimation by the clinician.
  * Demographics and disease-related information (i.e. age, sex, race, age at disease onset, disease duration)
  * Review of your medical records
  Interventions: Genetic: All Participants

INTERVENTIONS:
Genetic: All Participants — If you decide to participate in this study, we will collect 1 tablespoon (15 milliliters) of blood during the first/screening visit in order to extract your DNA.

SUMMARY:
Spinocerebellar ataxias (SCA) are genetic neurological diseases that cause imbalance, poor coordination, and speech difficulties. There are different kinds of SCA and this study will focus on types 1, 2,3, and 6 (SCA 1, SCA 2, SCA 3 , also known as Machado-Joseph disease and SCA 6). The diseases are rare, slowly progressive, cause increasingly severe neurological difficulties and are variable across and within genotypes. The purpose of this research study is to bring together a group of experts in the field of SCA for the purpose of learning more about the disease.

The research questions are:

1. How does your disease progress over time?
2. What are the best ways to measure the progression?
3. Do some genes, other than the gene that is abnormal in your disease, have any effect on the way the disease behaves?

This is a nationwide study and we expect that 800 patients will participate all over the USA. The participants will be in the study for an indeterminate period of time. Study visits will be done every 6 or 12 months depending on the participating site.

DETAILED DESCRIPTION:
If you decide to participate in this study, we will collect 1 tablespoon (15 milliliters) of blood during the first/screening visit in order to extract your DNA. The sample will be sent to the research laboratory of Dr Stefan Pulst at the University of Utah for the study of genetic factors that modify the course of your disease.

As part of this study, we would like to put some of your blood in a tissue repository. Submission of your sample to the repository may give scientists valuable research material that can help them to develop new diagnostic tests, new treatments, and new ways to prevent diseases. Scientists will not use your sample, or material isolated from it, for commercial products or services. Your blood will be kept by Dr. Stefan Pulst.

Your sample will not have your name or other personal information linked to it. Your sample may be shared with researchers at the University of Utah and at other institutions. The only information we will keep with the sample is your age, what disease you have, the age at onset of your disease and the duration of the disease. The principal investigator at your site will be the only person who can link the sample to you. You can have your sample removed from the bank later by written request to your PI.

You do not have to participate in the genetic modifier study or the tissue repository to be in the remaining part of this study.

You will also be asked to complete several assessments that include questionnaires, motor function test, a neurological exam and a physical exam.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptomatic ataxic disease
* Definite molecular diagnosis of SCA 1, 2,3,or 6 either in the subject or another affected family member
* Willingness to participate in the study and ability to give informed consent.
* Age 6 years and above

Exclusion Criteria:

* Known recessive, X-linked and mitochondrial ataxias
* Exclusion of SCA 1, 2, 3 and 6 by previous DNA testing,
* A lack of willingness to participate in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Clinical Research Consortium for Spinocerebellar Ataxias (CRC-SCA) is seeking subjects to participate in a clinical research study of patients with SCA 1, 2 3 and 6.
  Potential participants should have symptoms of ataxia with a diagnosis of SCA 1,2,3 or 6 established by DNA tests either on the patient himself or herself or another affected family member and be between 6 and 80 years of age. In addition, patients who have ataxia with a dominant inheritance pattern but who do not yet know what type of SCA they have can also be screened for this project.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2024-05-19 (Estimated); Study Completion 2024-05-19 (Estimated)

PRIMARY OUTCOMES:
The disease's progression over time using clinical rating scales and timed performance measures. | Indefinitely (for as long as the study is open and you wish to participate)
Relation between the genetic modifiers and the age at onset of disease and disease progression rates. | Indefinitely (for as long as the study is open and you wish to participate)

SECONDARY OUTCOMES:
The effects of the disease on the Activities of Daily Living (ADL)in patients with Spinocerebellar Ataxias | indefinitely

CONTACTS AND LOCATIONS:
Overall Officials: S. Subramony, MD, Principal Investigator — University of Florida
Locations (12):
- United States (12):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Harvard University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: National Ataxia Foundation — http://www.ataxia.org/